CLINICAL TRIAL: NCT07153926
Title: Vibration Controlled Tissue Elastography Versus Iron Regulators as Diagnostic Tools for Hepatic Fibrosis - Iron Overload in Egyptian Children With Beta- Thalassemia
Brief Title: Elastography vs Iron Regulators in the Diagnosis of Hepatic Fibrosis- Iron Overload in Children With Beta- Thalassemia
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rania Mamdouh Elkafoury, Lecturer of Tropical medicine, Tanta University
Other Study IDs: 36264PR872/9/24
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Liver Fibrosis; Beta Thalassemia Major
Keywords: Fibroscan; Liver fibrosis; Iron overload; Beta- thalassemia
MeSH Terms: conditions — Liver Cirrhosis; beta-Thalassemia; Iron Overload

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- beta- thalassemia patients: 100 beta-thalassemia major children with iron overload aged 5 to 18 years, as indicated by serum ferritin levels more than 500 ng/mL.
  Interventions: Diagnostic Test: Serum ferritin; Diagnostic Test: Serum hepcidin

INTERVENTIONS:
Diagnostic Test: Serum ferritin — Serum ferritin is a protein that stores iron, and high serum ferritin levels can suggest iron overload, but are also a common indicator of other conditions like inflammation, liver disease, or metabolic syndrome.
Diagnostic Test: Serum hepcidin — Hepcidin hormone has been found to be a key regulator of iron homeostasis. It controls plasma iron levels by regulating two key steps in iron metabolism, namely digestive iron absorption in enterocytes and iron recycling in macrophages.
  Hepcidin is synthesized predominantly in the hepatocytes, which is physiologically increased by elevated serum iron level and decreased by erythropoietic activity. Recently, hepcidin has been used as a new marker for evaluation of liver fibrosis in patients with thalassemia major.

SUMMARY:
The goal of this cross-sectional observational study is to evaluate the accuracy of serum ferritin and serum hepcidin versus non-invasive scores in the diagnosis of liver fibrosis and iron overload in beta- thalassemia children.

Researchers will measure and correlate serum ferritin, hepcidin and hepcidin/ferritin ratio in beta- thalassemia children with liver fibrosis. Researchers will also evaluate the performance of serum ferritin, hepcidin and hepcidin/ferritin ratio, AST to platelet ratio index (APRI) score, and fibrosis-4 (FIB-4) score, for predicting significant fibrosis (>=F2).

Participants will undergo history-taking, clinical examination, laboratory investigations, serum ferritin, serum hepcidin, abdominal ultrasonography, and Fibroscan examination. The APRI, FIB-4, and hepcidin/ferritin ratio will be calculated. The performance of serum ferritin, hepcidin and hepcidin/ferritin ratio for predicting significant fibrosis will be compared versus other non-invasive scores.

ELIGIBILITY:
Inclusion Criteria:

* Children with ß-thalassemia major
* iron overload, as indicated by serum ferritin levels more than 500 ng/mL.

Exclusion Criteria:

* Pediatric patients with liver diseases (such as hepatitis).
* children with other types of chronic hemolytic anemia.
* other chronic systemic diseases (DM and Hypertension) or malignancy or heart diseases.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This cross-sectional observational study will be carried out on 100 children and adolescents who are pre-diagnosed patients with ß thalassemia major and iron overload. Patients will be enrolled from the Pediatric Gastroenterology, Hepatology & Endoscopy and Hematology Units, Tanta University Hospital, Egypt. Fibroscan will be done in the Tropical Medicine and Infectious Diseases Department, Tanta University Hospital, Egypt. The start of research will begin in September 2024 and will end in December 2024.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
measuring hepcidin level (nanogram/ml) for predicting iron overload | through study completion, an average 6 months
measuring ferritin level (nanogram/ml) for predicting significant fibrosis | through study completion, an average 6 months
measuring hepcidin level (nanogram/ml) for predicting significant fibrosis | through study completion, an average of 6 months

SECONDARY OUTCOMES:
comparing serum ferritin versus non-invasive scores for significant fibrosis | through study completion, an average of 6 months
comparing serum hepcidin versus non-invasive scores for significant fibrosis | through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Gharbyea, Egypt